CLINICAL TRIAL: NCT00845559
Title: The Effects of Exenatide on Post-Prandial Glucose Excursions and Vascular Health in Obese/Pre-Diabetic Young Adults
Brief Title: The Effects of Exenatide on Post-Meal Sugar Peaks and Vascular Health in Obese/Pre-Diabetic Young Adults
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0801003390
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Obesity; Insulin Resistance; Impaired Glucose Tolerance; Cardiovascular Disease
Keywords: Childhood Obesity; Insulin resistance; Impaired Glucose Tolerance; Cardiovascular Disease; Type 2 Diabetes Mellitus; Continuous Glucose Monitoring (CGMS); Exenatide; Oral Glucose Tolerance Test
MeSH Terms: conditions — Obesity; Insulin Resistance; Glucose Intolerance; Cardiovascular Diseases; Pediatric Obesity; Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): Subjects randomized to treatment will receive a four month supply of exenatide.
  Interventions: Drug: Exenatide
- No Treatment (No Intervention)

INTERVENTIONS:
Drug: Exenatide — Subjects randomized to treatment will receive a four month supply of exenatide and will be taught how to administer subcutaneous injections with their exenatide pen and instructed on the following dosing schedule: exenatide - 5 μg twice a day for 7 days, followed by exenatide 10 μg twice a day for the remainder of the four month supply.
  Other Names: Byetta
  Arms: Exenatide

SUMMARY:
The primary aim of this study is to evaluate the effect of exenatide on daily glycemic excursions obtained by continuous glucose monitoring system (CGMS). The CGMS summary parameters that we are most interested in include:

* The percent of glucose values above 140 mg/dl and/or AUC of glucose values above 140 mg/dl
* AUC of glucose values over 100 mg/dl during three days
* Maximal meal-related glucose excursions
* Three-day mean glucose (including low readings - below 100 mg/dl)

Secondary Study Endpoints:

Secondary endpoints will include:

* glucose tolerance status as assessed by OGTT
* Vascular function scores as assessed by PAT, FMD and step test.
* Biochemical markers of vascular health, including inflammatory markers, markers of oxidative stress and microalbuminuria.
* Changes in BMI

DETAILED DESCRIPTION:
Obese insulin resistant adolescents with impaired glucose tolerance (IGT) or evidence of glucose excursions ≥ 140 mg/dl on CGMS will be enrolled in a two armed randomized, parallel group - open label study. There will also be a lean control group for baseline assessments only.

One arm will be exenatide the other arm will be no drug. Subjects will be stratified according to state of glucose tolerance. Stratification will also occur according to gender and family history of premature cardiovascular disease.

Obese adolescents age 16-25 years with a family history of type 2 diabetes, whom have completed or reached tanner IV stage of pubertal development and have normal or impaired oral glucose tolerance. Obese adolescents age 13-15 with a family history of type 2 diabetes, whom have completed or reached tanner III stage of pubertal development and have impaired oral glucose tolerance with a 2-hour glucose of 180-199 mg/dl will also be invited to participate. For cardiovascular assessment only age matched lean control subjects without diabetes will be recruited.

Obese subjects will have a baseline and post intervention oral glucose tolerance test (OGTT), screening labs (liver/kidney functions, lipid profile, thyroid function tests, CBC, metabolic and cardiovascular laboratory parameters -- such as inflammatory cytokines and pro-thrombotic factors), wear a CGMS for 3-days on 3 separate occasions (baseline, 2-month and 4-month), have a standardized snack once during each CGMS session, collect urine samples for microalbumin and have vascular tests (PAT, FMD and exercise step test) done at baseline and post intervention.

Subjects randomized to treatment will undergo a four month intervention with exenatide on the following dosing schedule: exenatide - 5 μg twice a day for 7 days, followed by exenatide 10 μg twice a day for the remainder of the four month intervention.

Lean Control Subjects:

As for obese subjects, lean subjects will be asked to bring in first morning voids for testing of microalbuminuria. They will also have endothelial function tests (PAT, FMD and step test) as well as CGMS placement. A set of screening labs will also be drawn (fasting glucose, insulin, thyroid function and lipid profile will be drawn). Furthermore blood will be collected for analysis of novel cardiovascular parameters (such as inflammatory cytokines and pro-thrombotic factors). However lean subjects will not have an OGTT done and will not be offered drug intervention. The endothelial function testing in the lean controls will serve as control data for the vascular function testing in the obese children. The CGMS data of the lean controls will allow us to better interpret changes in the post-meal excursions seen in obese children after exenatide intervention. Similar to obese subjects, lean subjects will be instructed to take a standardized snack in the afternoon prior to returning for CGMS removal. The snack will be provided for them to take home at the end of their CGMS placement visit and will include two pop-tarts and an orange soda. Lean control subjects will wear the CGMS for three days. At the end of the monitoring period the subject will return for their CGMS removal visit.

ELIGIBILITY:
Obese subjects:

Major Inclusion Criteria:

* Obesity (BMI > 97%tile for age and sex matched normative data)
* Insulin resistance: fasting insulin> 25 mIU/ml
* Good general health, taking no medication on a chronic basis
* Age 16-25 yrs, late pubertal stage (girls: breast: Tanner stage IV to V, boys: testicular volume > 15 ml) or age 13-15 yrs (with a family history of type 2 diabetes, whom have completed or reached tanner stage III and have impaired oral glucose tolerance with a 2-hour glucose of 180-199 mg/dl)
* Girls who are sexually active must use adequate birth control methods (such as barrier method or oral contraception) and must have a negative pregnancy test
* Normal liver function tests

Major Exclusion Criteria:

* Hx of gallstones
* Elevated triglycerides >400 mg/dl
* Hx of alcohol use/ binge drinking
* Raynaud's syndrome
* Pregnancy or breastfeeding mothers
* Cigarette smokers
* Anemia (Hct < 35)
* Baseline creatinine > 1.0 mg
* Abnormal liver transaminases > 2.0 X the upper limit of normal
* Presence of endocrinopathies except for adequately treated hypothyroidism
* Presence or history of gastrointestinal disorders (inflammatory bowl disease, irritable bowl disease, hernia, ileus)
* Presence of significant chronic illness of any kind.
* Use of any drugs that might be expected to affect glucose tolerance, insulin resistance or weight gain, cardiovascular health.
* Psychiatric disorders
* History of substance abuse

Lean Control Subjects (only for cardiovascular studies and CGMS):

Inclusion Criteria:

* Lean (BMI < 85%tile for age and sex matched normative data)
* Fasting insulin <15 mIU/m
* Fasting glucose <100 mg/dll
* Excellent general health, having no acute or chronic health problems and taking no current medications
* Age 13-25 yrs, in puberty (age matched with obese subjects)
* Girls who are sexually active must use adequate birth control methods (such as barrier method or oral contraception) and must have a negative pregnancy test

Exclusion Criteria:

* Raynaud's syndrome
* Pregnancy or breastfeeding mothers
* Cigarette smokers
* Psychiatric disorders
* History of substance abuse
* First degree relative with either T1DM or T2DM
* Presence of acanthosis nigricans

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Whether treatment with exenatide attenuates post-prandial glycemic excursions as assessed by oral glucose tolerance testing (OGTT) and continuous monitoring system (CGMS) technology. | OGTT (Pre- and post-intervention), CGMS (Pre-intervention, 2-months and post-intervention)

SECONDARY OUTCOMES:
Cardiovascular risk parameters will be assessed via flow mediated vasodilation, peripheral arterial tonometry, a self-paced step test and biochemical markers of vascular health. | Pre- (baseline) and post- (4-months) intervention
Change in body mass index (BMI). | Pre-intervention, 2-month and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tania S Burgert, MD, Principal Investigator — Yale University